CLINICAL TRIAL: NCT00172874
Title: Cross-Cultural Validity of EDI-1 Among Clinical and Non-Clinical Taiwanese Population
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Mei-Chih Tseng/Attending psychiatrist, National Taiwan University Hospital
Other Study IDs: 9461700313; NSC-89-2413-H002-016
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Eating Disorders
Keywords: cross-cultural,; eating disorders,; EDI,; psychometrics
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to understand the clinical characteristics of Taiwanese eating disorders as well as establishment of the psychometric properties of eating disorder-related questionnaires (EDI and BITE).

DETAILED DESCRIPTION:
The study subjects include three group of population: 1st group is non-clinical nursing college students (N=800); 2nd group is clinical eating disorder patients (N=600) and 3rd group is age-, sex-matched clinical non-eating disorder patients (N=600). Clinical patients are screened by eating disorder module of the SCID and are grouped into eating disorder or non-eating disorder group. After written informed consent, eating disorder patients will receive clinical assessments which included important clinical characteristics and psychopathology of eating disorders by experienced senior psychiatrists. All clinical patients are asked to complete the self-rating scales which included eating and general psychological functioning questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patients with eating disorders,
* patients with non-eating disorders,
* nursing school students

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinical patients with eating disorders, other psychiatric disorders, and students
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 1998-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chih Tseng, MD, Principal Investigator — National Taiwan Univetsity Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan